CLINICAL TRIAL: NCT00578942
Title: Allogeneic Non-myeloablative Stem Cell Transplantation Utilizing Matched Family Member Stem Cells Purged Using Campath-1H
Brief Title: Allo Non-myeloablative SCT Utilizing Matched Family Member Stem Cells Purged Using Campath
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: David Rizzieri, MD (Other)
Collaborators: Miltenyi Biomedicine GmbH (Industry)
Responsible Party: Sponsor-Investigator, David Rizzieri, MD, Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00008380
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Results first posted 2014-05-23 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-05

CONDITIONS: Lymphoma; Myeloma; Leukemia; Myelodysplasia; Solid Tumors
Keywords: Allogeneic Stem Cell Transplantation, Campath, HLA-Matched
MeSH Terms: conditions — Lymphoma; Neoplasms, Plasma Cell; Leukemia; Anemia, Refractory, with Excess of Blasts

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Campath Purged Non-myeloablative ASCT (Experimental): Campath Purged Non-myeloablative Allo Stem Cell Transplant (ASCT) in lymphoma, myeloma, or marrow failure: leukemia or myelodysplasia; and solid tumors
  Interventions: Drug: Campath Purged Non-myeloablative ASCT

INTERVENTIONS:
Drug: Campath Purged Non-myeloablative ASCT — Preparative regimen: Begins on day -5 and consist of 4 days of daily fludarabine at 30 mg/m2/d infused over 30 minutes, cyclophosphamide 500 mg/m2/d infused over 1 hour, 5 days of Campath-1H at 20 mg/d in 250 ml of D5 normal saline or normal saline infused over 3 hours.
  Subject Evaluation will occur 2-3 times per week by physical exam for toxicity through day 45.
  Other Names: Allogeneic Stem Cell Transplant (ASCT)

SUMMARY:
Allogeneic transplantation is used to treat many malignant and non-malignant diseases, though the potential toxicities of the procedure remain high. We and others have shown that a less toxic preparative regimen allows reliable allogeneic engraftment for allogeneic transplantation.

The primary purpose of this treatment trial is to follow subjects undergoing allogeneic transplantation for long term outcomes. The regimen used has been tested in our prior phase I / II trial which has completed accrual. The issues of engraftment and rate of graft versus host disease have been answered and our success has led to this regimen being a standard approach for less toxic allogeneic therapy.

DETAILED DESCRIPTION:
Allogeneic bone marrow transplantation may cure or ameliorate illnesses of many types; however the toxicity of the procedure limits its broad applicability. Hematologic malignancies of all types have shown responses. Those with marrow failure, such as aplasia, and hemoglobinopathies have further shown responses in multiple trials as well. Even patients with certain solid tumors, such as breast, renal cell, and melanoma have shown partial or complete responses to allogeneic therapy. The limiting effect of the historical methods of aggressive induction for allogeneic therapy were extremely toxic, requiring limiting those offered allogeneic therapy to the healthiest of the ill patients. Work over the last decade has shown that less toxic agents targeting the immune system effectively allowed engraftment with less effects on the patient's liver, lungs, and other vital organs. We and others have completed multiple trials showing the effective use of these less toxic, non-myeloablative, regimens for allogeneic therapy. Trials with fludarabine and cyclophosphamide at standard doses (patients are not ablated and recover blood counts in 2 weeks) allow for 80% of patients to engraft donor cells. Some groups have added low doses of radiation to this combination, with 80-100% allogeneic engraftment. The lessened toxicity of this approach has been confirmed in multiple studies, including our own data with the specific schema in this treatment plan reviewed below. Phase I results with this combination: Our group has combined the above combination of fludarabine and cyclophosphamide with the antibody CAMPATH 1H. This antibody is given to the patient to purge the immune system and prevent rejection. It also purges the T cells in the donated stem cells to minimize graft versus host disease (GVHD). This approach has been proven successful in multiple trials using standard more toxic ablative procedures. Our approach over the last 3 years has been very successful using this antibody with the less toxic non-myeloablative procedure and our trials have completed. We have presented our preliminary results, with data on long term follow up for outcomes being collected. We have shown that 100% of patients with a malignancy or marrow failure treated with this regimen in our early phase trial engrafted donor cells. There was only an 8% severe GVHD risk, though the risk for infection remains high with a risk of fungal and viral infection about 5% each. Despite working with older, more infirmed patients, only 3/40 patients died within the first 100 days from therapy. Similar approaches on matched unrelated donors have been reported by other groups as well. As the phase I feasibility trial is complete and the outcomes encouraging, this protocol will follow the same general treatment plan and allow further information to be gained for long term follow up of subjects treated with this approach.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have their pathology reviewed and the diagnosis confirmed.
* Performance status must be Cancer and Leukemia Group B (CALGB) performance score 0, 1, or 2
* Subjects must have a 6/6 Human leukocyte antigen (HLA)-matched related donor who is evaluated and deemed able to provide peripheral blood progenitor cells (PBPC) and/or marrow by the transplant team.
* HIV antibody negative.
* Subjects must test negative serum beta-human chorionic gonadotropin (HCG) and must agree to use some form of adequate birth control during the periods they receive chemotherapy and any post-chemotherapy medications related to the transplant.
* Subjects must be >/=17 years of age
* Subjects must also have a resting multigated acquisition (MUGA) and/or ECHO and pulmonary function test (PFT) with diffusion capacity of lung (DLCO) performed before transplant and found to be acceptable according to the treating institution's guidelines. The required minimum standards include MUGA and/or ECHO showing an ejection fraction (EF) of 40% and PFTs showing DLCO of 40%. Those with an EF 40-50%, undergo cardiac evaluation and consultation. Also, those with DLCO 40-50%, undergo pulmonary evaluation and consultation.
* Specific populations for each disease category:

A) Hematologic malignancies Those with high risk or relapsed hematologic malignancy (including myeloid and lymphoid leukemias and lymphomas, myeloma or myelomatous like diseases, myeloproliferative disease, myelodysplasia). Those with good risk disease (first remission acute myeloid leukemia (AML) with inv 16 M4 Eos, M3 AML with t(15;17); or t(8;21) in first remission are not eligible).

B) Bone marrow failure

1. Those specifically with idiopathic or secondary moderate, severe or very severe aplastic anemia (idiopathic or secondary) according to the accepted 'Camitta criteria' would be candidates.
2. Those with diseases known to lead to severe marrow failure are eligible as well. These include those with myelofibrosis or paroxysmal nocturnal hemoglobinuria (PNH).

C) Solid Tumors Subjects must have had a biopsy confirming disease recurrence (metastases) at some point in their history, unless the patient presented with metastatic disease, in which case the initial primary site biopsy is adequate.

1. Subjects with renal cell cancer, or melanoma will be eligible for this approach at this time. Subjects will have had documented metastatic disease at some time in the past. Subjects who are in remission or with residual disease after prior therapy for their metastatic disease are eligible, as there is no accepted cure for these patients with metastatic disease.
2. Breast Cancer- Subjects will have had documented metastatic disease at some time in the past. Subjects who are in remission or with residual disease after prior therapy for their metastatic disease are eligible. Subjects must have failed at least one chemotherapy regimen for their metastatic disease and 1 hormonal agent if they are receptor positive.

Exclusion Criteria:

1. pregnant or lactating women,
2. patients with other major medical or psychiatric illnesses which the treating physician feels could seriously compromise tolerance to this protocol, and
3. Leukemia patients in first remission with good risk cytogenetics for leukemia [t(15;17); t(8,22)]

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2005-05; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Rizzieri, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Health Systems, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was opened and first consent obtained on 9/11/2002 and was closed to accrual on 2/18/2008 as enrollment goal was met. Recruitment took place at Duke hospital in the Bone Marrow Transplant clinic during time of clinical appointments in a private location. Follow up for survival was discontinued in April 2013.
Pre-assignment Details: Prior to selecting a donor: donor and subjects had history and physical exam, labs and chest x-ray performed per program and FACT requirements. Female donors should have a negative pregnancy test. Subjects also had bone marrow aspirate/biopsy. Subjects were premedicated with Benadryl and acetaminophen.
Groups:
- Campath Purged Non-myeloablative ASCT: Campath Purged Non-myeloablative Allo Stem Cell Transplant (ASCT) in lymphoma, myeloma, or marrow failure: leukemia or myelodysplasia; and solid tumors
  Preparative regimen: Begins on day -5 and consist of 4 days of daily fludarabine at 30 mg/m2/d infused over 30 minutes, cyclophosphamide 500 mg/m2/d infused over 1 hour, 5 days of Campath-1H at 20 mg/d in 250 ml of D5 normal saline or normal saline infused over 3 hours.
  Subject Evaluation will occur 2-3 times per week by physical exam for toxicity through day 45.
Period: Overall Study
Arm/Group | Campath Purged Non-myeloablative ASCT
Started | 48
Completed | 47
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Cohort of subjects who actually received at least 1 donor lymphocyte infusion (DLI).
  DLI dosages thus ranged from 1×104 CD3+ cells/kg to 3.27 ×108 CD3+ cells/kg.
Groups:
- Campath Purged Non-myeloablative ASCT: Campath Purged Non-myeloablative Allo Stem Cell Transplant (ASCT) in lymphoma, myeloma, or marrow failure: leukemia or myelodysplasia; and solid tumors
  Preparative regimen: Begins on day -5 and consist of 4 days of daily fludarabine at 30 mg/m2/d infused over 30 minutes, cyclophosphamide 500 mg/m2/d infused over 1 hour, 5 days of Campath-1H at 20 mg/d in 250 ml of D5 normal saline or normal saline infused over 3 hours.
  Patient Evaluation will occur 2-3 times per week by physical exam for toxicity through day 45.
Arm/Group | Campath Purged Non-myeloablative ASCT
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 41
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 42
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 47
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 48

OUTCOME MEASURES:

1. Primary Outcome: Toxicity
Description: Acute graft versus host disease (GVHD) was graded according to the consensus criteria and NCI common terminology criteria for adverse events (CTCAE) v2.0 or 3.0 was used for all other toxicities. Recognizing that acute GVHD pathology in the nonablative and donor lymphocyte infusion (DLI) setting may occur late, we tabulated skin, gut and liver toxicity consistent with acute GVHD (aGVHD) at anytime in the year following the infusion as aGVHD. Toxicities were formally recorded for all patients twice weekly for the first 100 days, at each follow up visit, and as needed intercurrently.
Time Frame: 1 year
Population: Cohort of subjects who received >/=1 donor lymphocyte infusion (DLI). DLI doses thus ranged from 1×104 CD3+ cells/kg to 3.27 ×108 CD3+ cells/kg.Subjects were grouped into 4 categories within the range of cell doses delivered and were considered evaluable from the day of first donor lymphocyte (DLI) infusion. Results are not exclusive.
Measure: Number; unit: participants
Groups:
- Campath Purged Non-myeloablative ASCT: Campath Purged Non-myeloablative Allo Stem Cell Transplant (ASCT) in lymphoma, myeloma, or marrow failure: leukemia or myelodysplasia; and solid tumors
  Donor will receive Granulocyte colony-stimulating factor (G-CSF) 8 mcg/kg/d subcutaneously twice daily (dose will be rounded to the nearest whole vial size), Granulocyte-macrophage colony-stimulating factor (GM-CSF) 15 mcg/kg/d subcutaneous or similar growth factor for donor mobilization. Donors will receive at least 3-6 doses of daily growth factor until adequate cells are mobilized.
  Preparative regimen: Begins on day -5 and consist of 4 days of daily fludarabine at 30 mg/m2/d infused over 30 minutes, cyclophosphamide 500 mg/m2/d infused over 1 hour, 5 days of Campath-1H at 20 mg/d in 250 ml of D5 normal saline or normal saline infused over 3 hours.
  Subject Evaluation will occur 2-3 times per week by physical exam for toxicity through day 45.
Arm/Group | Campath Purged Non-myeloablative ASCT
Number analyzed (Participants) | 48
participants
  acute Graft versus Host Disease | 21
  Death | 25

2. Primary Outcome: Overall Survival (OS)
Description: Estimate overall survival rates in subjects treated with a non-myeloablative preparative regimen followed by matched related allogeneic stem cells for allogeneic transplantation.
Time Frame: Up to 12 years; participants were followed for the duration of the study, an average of 8 years
Population: Subjects who completed CAMPATH regimen + 45 days, until disease progression, or death. One participant who was lost to follow-up after 14 months was not included. Participants were followed for the duration of the study, an average of 8 years.
Measure: Mean (Full Range); unit: months alive post-infusion
Arm/Group | Campath Purged Non-myeloablative ASCT
Number analyzed (Participants) | 47
months alive post-infusion | 32 [2 to 123]

3. Secondary Outcome: Response
Description: Response Assessment included physical exam and evaluation of peripheral blood and bone marrow. There's no widely accepted criteria for response other than complete response (CR).
  CR for malignant hematologic diseases is met if all the following are met for >/= 1 month:
  1. absence of pathologic lymphadenopathy by physical and radiographic exam
  2. absence of constitutional symptoms due to disease
  3. Polymorphonuclear leukocyte count > 1,500/uL; platelet count >50,000/uL; and hemoglobin >10.0 g/dL
  4. bone marrow aspirate/biopsy done after (a) through (c) have been met, >/= 30% cellularity and an absence of abnormal lymphoid nodules or cells by flow cytometry, cytogenetics, etc.
  5. molecular markers of disease must be negative by polymerase chain reaction, Fluorescence in situ hybridization, cytogenetics etc.
  CR for solid tumors requires complete resolution of disease on physical exam and radiographs. CR for marrow failure is normal white cell, platelet and hematocrit values.
Time Frame: 1 year
Population: Cohort of subjects on the study who actually received >/=1 donor lymphocyte infusion (DLI). DLI doses ranged from 1×104 CD3+ cells/kg to 3.27 ×108 CD3+ cells/kg. Subjects were considered for a second and third DLI 8 weeks apart if they did not have >grade 2 toxicity from the initial DLI, donor availability, and insurance approved the infusion.
Measure: Number; unit: participants
Arm/Group | Campath Purged Non-myeloablative ASCT
Number analyzed (Participants) | 48
participants | 18

ADVERSE EVENTS:
Time Frame: Toxicities were formally recorded for all patients twice weekly for the first 100 days, at each follow up visit, and as needed intercurrently, up to 10 years
Description: NCI Common Terminology Criteria for Adverse Events version 3 was used to grade toxicities. The drug manufacturer, Berlex, required the reporting of all Serious Adverse Events associated with the study to Berlex Global Medical Safety Surveillance Group.
Arm/Group | Campath Purged Non-myeloablative ASCT
Serious Adverse Events (participants affected / at risk) | 36/48
Other Adverse Events (participants affected / at risk) | 48/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Campath Purged Non-myeloablative ASCT (N=48)
Death (General disorders) | 36 (36)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 (1) — e.g. thrombotic thrombocytopenic purpura [TTP] or hemolytic uremic syndrome [HUS]
Hemorrhage (Vascular disorders) | 5 (6)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Campath Purged Non-myeloablative ASCT (N=48)
Allergic reaction / hypersensitivity (Immune system disorders) | 2 (2)
Hypotension (Vascular disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 8 (9)
Vomiting (Gastrointestinal disorders) | 4 (4)
Febrile neutropenia (Blood and lymphatic system disorders) | 16 (21) — fever of unknown origin without clinically or microbiologically documented infection)(ANC <1.0 x 10e9/L, fever >=38.5 degrees C
Creatinine (Investigations) | 3 (4)
Neuropathy: motor (Nervous system disorders) | 1 (2)
Neuropathy: sensory (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) — shortness of breath
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 (6) — lack of oxygen
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Failure to engraft (Gastrointestinal disorders) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 2 (2)
Cardiac Left Ventricular Function (Cardiac disorders) | 2 (3)
Infection with Grade 3 or 4 neutrophils (Infections and infestations) | 12 (16)
Infection with normal ANC or Grade 1/2 neutrophils (Infections and infestations) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes